CLINICAL TRIAL: NCT02286765
Title: Optimization of the Ulthera® System for Treating Axillary Hyperhidrosis
Brief Title: Ulthera® System for Treating Axillary Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ULT-126
Record Dates: First submitted 2014-11-05; First posted 2014-11-10 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-06

CONDITIONS: Primary Axillary Hyperhidrosis
Keywords: Ulthera System; Ultherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Subjects receiving Ulthera System treatment in a 3 x 4 grid, 12 treatment squares, 60 lines of treatment per square, at one treatment depth (2.0mm), at 0.30 J of energy
  Interventions: Device: Ulthera System treatment
- Group B (Active Comparator): Subjects receiving Ulthera System treatment in a 3 x 4 grid, 12 treatment squares, 40 lines of treatment per square, at one treatment depth (2.0mm), at 0.30 J of energy
  Interventions: Device: Ulthera System treatment

INTERVENTIONS:
Device: Ulthera System treatment — Micro-focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy

SUMMARY:
Up to 20 enrolled subjects will be treated. Subjects will receive two Ulthera® treatments on the axillas provided 30 days apart. Follow-up visits will occur at 7, 30, 90 and 180 days following the last treatment.

Protocol amendment: The study was expanded to enroll an additional 20 subjects into Group A.

DETAILED DESCRIPTION:
This study is a prospective, single-center, randomized clinical trial. Up to 20 subjects who are naïve to Ultherapy for treatment of hyperhidrosis will be enrolled and treated at a 2.0mm depth at two different treatment densities (Group A and Group B).

Group A will include up to 10 treated subjects. Subjects receiving treatment in a 3 x 4 grid, 12 treatment squares, 60 lines of treatment per square, at one treatment depth (2.0mm), at 0.30 J of energy.

Group B will include up to 10 treated subjects. Subjects receiving treatment in a 3 x 4 grid, 12 treatment squares, 40 lines of treatment per square, at one treatment depth (2.0mm), at 0.30 J of energy.

Gravimetric sweat production measures and starch iodine tests will be completed at baseline, treatment visit #2, and at all follow-ups for all study groups. Digital images of the starch iodine test will be obtained. Hyperhidrosis Disease Severity Scale (HDSS) scores will be obtained at baseline, each treatment visit, and at all follow-ups for all study groups.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-75 years.
* Subject in good health.
* Diagnosis of bilateral axillary hyperhidrosis refractory to previous topical therapies.
* At least 50 mg of spontaneous resting axillary sweat production in each axilla measured gravimetrically at room temperature/humidity (20 - 25.6°C/20-80%) over a period of 5 minutes. (Patients should be at rest for at least 30 minutes after physical exercise including walking.)
* HDSS score of 3 or 4. An attempt will be made to approximate an equal number of scores 3 and 4.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the Screening Visit and be willing and able to use an acceptable method of birth control (e.g. barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following conditions is documented on the medical history:

  1. Postmenopausal for at least 12 months prior to study;
  2. Without a uterus and/or both ovaries; or
  3. Bilateral tubal ligation at least six months prior to study enrollment.
* Absence of physical or psychological conditions unacceptable to the investigator.
* Willingness to refrain from use of aspirin, Ibuprofen, Naproxen or any other NSAID, and Vitamin E in the 2 weeks prior to each study treatment .
* Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure.

Exclusion Criteria:

* Dermal disorder including infection at anticipated treatment sites in either axilla.
* Previous botulinum toxin treatment of the axilla in the past year.
* Expected use of botulinum toxin for the treatment of any other disease during the study period.
* Known allergy to starch powder, iodine, lidocaine, or epinephrine.
* Secondary hyperhidrosis, for example, hyperhidrosis that is secondary to other underlying diseases including hyperthyroidism, lymphoma and malaria.
* Previous surgical treatment of hyperhidrosis including sympathectomy, surgical debulking of the sweat glands, subcutaneous tissue curettage and ultrasonic surgery.
* Unwillingness to wash off deodorants and abstain use 72 hours prior to treatments or assessments.
* Subjects with a history of a bleeding disorder
* Active implants (e.g., pacemakers or defibrillators), or metallic implants in the treatment areas.)
* Use of cholinomimetics, anticholinergics, or any oral herbal medicine treatments for hyperhidrosis.
* Inability to withhold use of antiperspirants and deodorants, or any other topical treatments for hyperhidrosis within 72 hours prior to study treatments and assessments.
* Unwillingness for complete shaving or removal of underarm hair within 12 hours prior to study treatments and follow-up visits.
* Women who are pregnant, lactating, possibly pregnant or planning a pregnancy during the study period.
* Inability to understand the protocol or to give informed consent.
* History of chronic drug or alcohol abuse.
* History of autoimmune disease.
* Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
* Subjects who anticipate the need for surgery or overnight hospitalization during the study.
* Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
* Concurrent enrollment in any study involving the use of investigational devices or drugs.
* Use of antiplatelet agents / Anticoagulants (Coumadin, Heparin, Plavix) in the past 6 weeks;
* Psychiatric drugs that in the investigators opinion would impair the subject from understanding the protocol requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
HDSS score reduction | Day 30 post-treatment #2
  HDSS score reduction from a 3 or 4 at baseline to a 1 or 2 at 30 days post-treatment #2.

SECONDARY OUTCOMES:
Sweat production by gravimetric measure | 7 Days post-treatment #2
  Reduction in spontaneous axillary sweat production assessed by a gravimetric method, as measured by a 50% reduction or more compared to baseline.
  • Gravimetric method is performed by drying the surface of the skin, then applying a pre-weighed filter paper to the axilla for a period of time measured by a stopwatch. The paper is then weighed and the rate of sweat production is calculated in mg/min.
Sweat production by gravimetric measure | 90 Days post-treatment #2
  Reduction in spontaneous axillary sweat production assessed by a gravimetric method, as measured by a 50% reduction or more compared to baseline.
  • Gravimetric method is performed by drying the surface of the skin, then applying a pre-weighed filter paper to the axilla for a period of time measured by a stopwatch. The paper is then weighed and the rate of sweat production is calculated in mg/min.
Sweat production by gravimetric measure | 30 Days post-treatment #2
  Reduction in spontaneous axillary sweat production assessed by a gravimetric method, as measured by a 50% reduction or more compared to baseline.
  • Gravimetric method is performed by drying the surface of the skin, then applying a pre-weighed filter paper to the axilla for a period of time measured by a stopwatch. The paper is then weighed and the rate of sweat production is calculated in mg/min.
Sweat production by gravimetric measure | 180 Days post-treatment #2
  Reduction in spontaneous axillary sweat production assessed by a gravimetric method, as measured by a 50% reduction or more compared to baseline.
  • Gravimetric method is performed by drying the surface of the skin, then applying a pre-weighed filter paper to the axilla for a period of time measured by a stopwatch. The paper is then weighed and the rate of sweat production is calculated in mg/min.
HDSS score reduction | 90 Days post-treatment #2
  HDSS score reduction from a 3 or 4 to a 1 or 2 at 90 days post treatment #2.
Starch iodine test | 7 Days post-treatment #2
  Starch iodine test to assess area of efficacy with digital images.
  • Starch Iodine test is performed by applying an iodine solution to the sweaty area. After it dries, starch is sprinkled on the area. The starch-iodine combination turns a dark blue color wherever excess sweat is present. Digital images of the starch iodine test will be obtained.
Starch iodine test | 30 Days post-treatment #2
  Starch iodine test to assess area of efficacy with digital images.
  • Starch Iodine test is performed by applying an iodine solution to the sweaty area. After it dries, starch is sprinkled on the area. The starch-iodine combination turns a dark blue color wherever excess sweat is present. Digital images of the starch iodine test will be obtained.
Starch iodine test | 90 Days post-treatment #2
  Starch iodine test to assess area of efficacy with digital images.
  • Starch Iodine test is performed by applying an iodine solution to the sweaty area. After it dries, starch is sprinkled on the area. The starch-iodine combination turns a dark blue color wherever excess sweat is present. Digital images of the starch iodine test will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Larson, MBA, Study Director — Ulthera, Inc
Locations (1):
- Saint Louis University Dermatology, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No